CLINICAL TRIAL: NCT07222969
Title: An Open-label, Dose-escalation and Dose-expansion Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic (PK) Characteristics, and Preliminary Efficacy of VIB305 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study to Evaluate the Safety of VIB305 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vibrant Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIB305-001
Record Dates: First submitted 2025-10-22; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- VIB305 for Injection in Cohort 1 (Experimental): VIB305 for Injection does in Cohort 1 according to protocol
  Interventions: Drug: VIB305 for Injection
- VIB305 for Injection in Cohort 2 (Experimental): VIB305 for Injection does in Cohort 2 according to protocol
  Interventions: Drug: VIB305 for Injection
- VIB305 for Injection in Cohort 3 (Experimental): VIB305 for Injection does in Cohort 3 according to protocol
  Interventions: Drug: VIB305 for Injection
- VIB305 for Injection in Cohort 4 (Experimental): VIB305 for Injection does in Cohort 4 according to protocol
  Interventions: Drug: VIB305 for Injection
- VIB305 for Injection in Cohort 5 (Experimental): VIB305 for Injection does in Cohort 5 according to protocol
  Interventions: Drug: VIB305 for Injection
- VIB305 for Injection in Cohort 6 (Experimental): VIB305 for Injection does in Cohort 6 according to protocol
  Interventions: Drug: VIB305 for Injection

INTERVENTIONS:
Drug: VIB305 for Injection — Intravenous infusion: once every week, each treatment cycle is 3 weeks.

SUMMARY:
This clinical trial is an open-label, single-arm, non-randomized, dose-escalation and dose-expansion study targeting subjects with unresectable, advanced, malignant solid tumors who have failed or are unsuitable for standard treatments or refused the existing treatments.

This study is divided into a dose-escalation phase (Phase I) and a dose-expansion phase (Phase II). Phase I (dose escalation) is designed to preliminarily evaluate the safety and tolerability of VIB305 in advanced solid tumors, to determine the nature and incidence of dose-limiting toxicities (DLTs), and thereby to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). Based on the findings from the Phase I portion for evaluation in the Phase II portion. Phase II (dose expansion) will enroll additional cohorts to further assess the safety and tolerability, PK profile, preliminary antitumor activity and immunogenicity of VIB305 in specific tumor types (selected based on all available data).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, male or female.
2. Subjects with histologically or cytologically confirmed advanced solid tumors that are unresectable, who are refractory to or intolerant of or refuse all existing therapy(ies) known to provide clinical benefit for their condition.
3. At least one measurable lesion as assessed by RECIST 1.1.
4. ECOG performance status score of 0-1.
5. Estimated survival time of more than 3 months.
6. Adequate organ function.
7. Females of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to first administration of the investigational drug. Females of childbearing potential must agree to abstain or use highly effective contraception from the time of signing informed consent form until 6 months after their last dose of the investigational drug.
8. Male subjects of reproductive capacity must agree to use effective contraception from the time of signing informed consent form until 6 months after their last dose of the investigational drug.
9. Subjects must be fully informed about this study before participation and must voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Receipt of chemotherapy, biotherapy, endocrine therapy, immunotherapy, or other systemic anti-tumor therapy within 4 weeks prior to first dose of investigational drug.
2. Receipt of radiotherapy within 4 weeks prior to initiation of study treatment, or history of radiation pneumonitis.
3. Receipt of any other investigational drugs not yet marketed within 4 weeks prior to first dose of investigational drug.
4. Receipt of major organ surgery or occurrence of significant trauma, or requirement for elective surgery during the study, within 4 weeks prior to first dose of investigational drug.
5. Use of systemic glucocorticoids or other immunosuppressive agents within 14 days prior to the first dose of investigational drug or anticipated need during the study.
6. Use of immunomodulatory agents, including but not limited to thymosin, interleukin-2, interferons, etc., within 14 days prior to first administration of investigational drug.
7. Receipt of live vaccine or attenuated live vaccine within 4 weeks prior to first use of investigational drug. Inactivated vaccines are permitted.
8. History of prior allogeneic bone marrow transplantation or organ transplantation.
9. Adverse reactions from prior anti-tumor therapy have not recovered to ≤ Grade 1 based on CTCAE v5.0.
10. Subjects with central nervous system (CNS) metastasis.
11. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to first dose.
12. Known history of human immunodeficiency virus (HIV) positivity or history of acquired immunodeficiency syndrome (AIDS).
13. Subjects with active hepatitis B virus (HBV) infection.
14. History of other malignancies within the past 5 years.
15. History of severe cardiovascular or cerebrovascular disease.
16. Clinically significant severe pulmonary dysfunction.
17. Subjects with active or recurrent autoimmune diseases, or a related history and high risk for recurrence, or subjects at high risk.
18. Subjects with ulcerative keratitis, acute keratitis, or progressive keratitis.
19. Subjects with severe skin diseases.
20. Known hypersensitivity or allergy to any component of the investigational drug.
21. Prior receipt of immunotherapy, with severe immune-related toxicity regardless of remission status, as determined by the investigator to be unsuitable for immunotherapy.
22. Clinically uncontrolled pericardial, pleural, or peritoneal effusions requiring repeated drainage.
23. Dementia or altered mental status that may impair understanding and provision of informed consent form.
24. Pregnant or lactating females.
25. Underlying conditions.
26. Prior receipt of treatment with T cell engager drugs containing CD3 monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
MTD and/or RP2D based on the incidence and nature of DLTs | At the end of Cycle 1 (each cycle is 21 days)
  Incidence of dose-limiting toxicities (DLTs)
Adverse events（AE） | From signed ICF to 30 days after the last drug administration
  Include SAEs, TEAEs

SECONDARY OUTCOMES:
The immunogenicity of VIB305 | Pre-dose of Cycle 1, Cycle 1 Day 15, pre-dose of Cycle 2, Cycle 2 Day 15, pre-dose of Cycle 3, Cycle 4 and following cycle(each cycle is 21 days) , 30 days after the last administration, 90 days after the last administration
  Specification and quantification of ADAs or NAb
Objective response rate (ORR) | From signed ICF to 30 days after the last drug administration
  The proportion of subjects who achieved a confirmed response of complete response (CR) or partial response [PR]
Duration of response (DOR) | From signed ICF to 30 days after the last drug administration
  The time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD)
Disease control rate(DCR) | From signed ICF to 30 days after the last drug administration
  The proportion of patients who achieved complete response (CR), partial response (PR), and stable lesion (SD) after tumor treatment and could maintain the minimum duration requirement
Progression-free survival (PFS) | From signed ICF to 30 days after the last drug administration
  The time from the date of enrollment to the earlier of the dates of the first objective documentation of radiographic PD based on RECIST version 1.1 or death due to any cause
The pharmacokinetics (PK) profile of VIB305（Maximum concentration (Cmax)） | Cycle 1(Day 1, Day 2, Day 4,Day 6, Day 8, Day 15), Cycle 2(Day 1,Day 2, Day 4,Day 6, Day 8), Cycle 3 Day 1 and following cycle Day 1, each cycle is 21 days
  Maximum concentration (Cmax)
The pharmacokinetics (PK) profile of VIB305（Time of Cmax (Tmax)） | Cycle 1(Day 1, Day 2, Day 4,Day 6, Day 8, Day 15), Cycle 2(Day 1,Day 2, Day 4,Day 6, Day 8), Cycle 3 Day 1 and following cycle Day 1, each cycle is 21 days
  Time of Cmax (Tmax)
The pharmacokinetics (PK) profile of VIB305（Area under the curve (AUC)） | Cycle 1(Day 1, Day 2, Day 4,Day 6, Day 8, Day 15), Cycle 2(Day 1,Day 2, Day 4,Day 6, Day 8), Cycle 3 Day 1 and following cycle Day 1, each cycle is 21 days
  Area under the curve (AUC)
The pharmacokinetics (PK) profile of VIB305（Terminal half-life (t½)） | Cycle 1(Day 1, Day 2, Day 4,Day 6, Day 8, Day 15), Cycle 2(Day 1,Day 2, Day 4,Day 6, Day 8), Cycle 3 Day 1 and following cycle Day 1, each cycle is 21 days
  Terminal half-life (t½)